CLINICAL TRIAL: NCT04551014
Title: Randomized Controlled Trial Investigating Use of Submucosal Injection of EverLift in Rates of Complete Resection of Nonpedunculated Polyps 4-9mm
Brief Title: Evaluation of EverLift in the Performance of Polypectomy for Polyps 4-9mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Shai Friedland, Professor in Gastroenterology & Hepatology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15766-2
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Colo-rectal Cancer; Polyp of Colon; Adenomatous Polyp of Colon
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- With EverLift (Experimental): Polypectomy performed for polyps 4-9mm with submucosal injection of EverLift.
  Interventions: Device: Use of EverLift
- Without EverLift (Experimental): Polypectomy performed for polyps 4-9mm without submucosal injection of EverLift.
  Interventions: Device: Without use of EverLift

INTERVENTIONS:
Device: Use of EverLift — Use of EverLift for submucosal injection prior to polypectomy
  Arms: With EverLift
Device: Without use of EverLift — Without use of EverLift for submucosal injection prior to polypectomy
  Arms: Without EverLift

SUMMARY:
The focus of the study is to evaluate impact of submucosal injection of EverLift in achieving complete resection during polypectomy of polyps 4-9mm during colonoscopy.

DETAILED DESCRIPTION:
The details of the proposed study are as follows:

1. Experimental group: using EverLift submucosal injection for polyps 4-9mm of the colon
2. Control group: not using EverLift submucosal injection for polyps 4-9mm of the colon
3. Methods:

   1. Colonoscopy will be performed in the same standard of care manner as if no study was taking place.
   2. If polyps 4-9mm are identified, the endoscopist is randomized to performing polypectomy with or without submucosal injection of EverLift.
   3. After removal of the polypectomy, two biopsies are performed at the margin of the polypectomy site to identify residual lesion.
   4. The polyp as well as well as the two biopsies are reviewed by a pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Polyps 4-9mm

Exclusion Criteria:

* Pregnant
* Inflammatory bowel disease
* Polyposis syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shai Friedland, MD, Principal Investigator — Stanford University
Locations (1):
- Veterans Affairs Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each polyp sized 4-9 mm underwent block randomization to being removed by cold snare polypectomy (CNP) with or without submucosal injection of EverLift™.
Units Other Than Participants: Polyps
Groups:
- Polypectomy With EverLift: Polypectomy performed for polyps 4-9mm with submucosal injection of EverLift.
- Polypectomy Without EverLift: Polypectomy performed for polyps 4-9mm without submucosal injection of EverLift.
Period: Overall Study
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
Started | 105; 142 Polyps | 109; 149 Polyps
Completed | 105; 142 Polyps | 109; 149 Polyps
Not Completed | 0; 0 Polyps | 0; 0 Polyps

BASELINE CHARACTERISTICS:
Units Other Than Participants: Polyps
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift | Total
Number analyzed (Participants) | 105 | 109 | 158
Number analyzed (Polyps) | 142 | 149 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 27 | 51
  >=65 years | 81 | 82 | 163
Sex/Gender, Customized [Number; unit: participants]
  Female | 3 | 2 | 3
  Male | 102 | 107 | 155
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 3 | 4
  African American | 10 | 12 | 16
  Hispanic | 13 | 16 | 21
  White | 75 | 74 | 109
  Other | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 105 | 109 | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of Polyps With Complete Resection
Description: The primary outcome measured is comparison of completeness of resection between the with EverLift and without EverLift groups.
Time Frame: 2 weeks
Population: Participants with polyps randomized the respective procedure are included in the analysis
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
Number analyzed (Participants) | 105 | 109
Number analyzed (Polyps) | 142 | 149
Polyps | 140 | 145
Statistical Analysis 1: Comparison: Polypectomy With EverLift vs Polypectomy Without EverLift; Test type: Non-Inferiority — For polypectomy without submucosal injection of EverLiftTM to be considered non-inferior, we calculated that 115 polyps were needed in each group to achieve an alpha value of 0.05, power of 90%, and non-inferiority margin of -10%; p = 0.424, t-test, 2 sided

2. Secondary Outcome: Time to Resection
Description: The time between the snare is introduced till the polyp is removed and retrieved will be compared between the with and without EverLift groups.
Time Frame: During the procedure
Population: Participants with polyps randomized the respective procedure are included in the analysis
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Polyps
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
Number analyzed (Participants) | 105 | 109
Number analyzed (Polyps) | 139 | 146
Seconds | 109.8 (56.0) | 38.8 (54.5)
Statistical Analysis 1: Comparison: Polypectomy With EverLift vs Polypectomy Without EverLift; Test type: Superiority; p < 0.0001, t-test, 2 sided — P-value of <0.05 was considered statistically significant

3. Secondary Outcome: Number of Polyps Requiring Multiple Snare Attempts to Achieve Complete Endoscopic Polypectomy.
Time Frame: During the procedure (up to 10 minutes)
Population: Participants with polyps randomized the respective procedure are included in the analysis
Measure: Count of Units; unit: Polyps
Units Other Than Participants: Polyps
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
Number analyzed (Participants) | 105 | 109
Number analyzed (Polyps) | 142 | 149
Polyps | 6 | 5
Statistical Analysis 1: Comparison: Polypectomy With EverLift vs Polypectomy Without EverLift; Test type: Superiority; p = 0.697, Chi-squared — P-value of <0.05 was considered statistically significant

4. Secondary Outcome: Number of Patients With Procedural Complications
Description: Procedural complications include perforation and immediate post-polypectomy bleeding, early post-polypectomy bleed (within 24 hours) and delayed post polypectomy bleed (between 24 hours and 30 days). Early post-polypectomy bleed and delayed post-polypectomy bleed is evaluated based on emergency room (ER) visit, inpatient stay, transfusion needed, repeat colonoscopy required, surgical intervention required, and mortality.
Time Frame: 4 weeks (from procedure through 30 day follow-up)
Population: Participants with polyps randomized the respective procedure are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
Number analyzed (Participants) | 105 | 109
Participants | 1 | 2

ADVERSE EVENTS:
Time Frame: 30 days
Description: Patients who had the respective procedure were considered at risk for that procedure.
Arm/Group | Polypectomy With EverLift | Polypectomy Without EverLift
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/109
Serious Adverse Events (participants affected / at risk) | 1/105 | 2/109
Other Adverse Events (participants affected / at risk) | 0/105 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polypectomy With EverLift (N=105) | Polypectomy Without EverLift (N=109)
Splenic artery thrombosis (Vascular disorders) | 1 | 1
Post-polypectomy bleeding (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04551014/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT04551014/SAP_001.pdf